CLINICAL TRIAL: NCT06604143
Title: Discovering the Potential for Motor Recovery in People Living With Stroke
Brief Title: Stroke Motor Recovery for the Hand and Fingers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); McGill University (Other)
Responsible Party: Principal Investigator, Joyce Chen, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 46065; G-23-0034937 (Other Grant/Funding Number: Heart and Stroke Foundation of Canada)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Motor system; Stroke rehabilitation; Magnetic resonance imaging; Kinematics; Music
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To keep the study fair and unbiased, the participants, principal investigator, and the people analyzing the data won't know which training method each participant is using. This means they will be "blinded" to the study groups. If participants knew why the study groups were chosen and which group they were in, it might affect their performance and the study results.
  However, the therapist delivering the piano training will know which method is being used. To reduce bias, this therapist won't be involved in analyzing the data or know the research goals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quality Training Group (Active Comparator)
  Interventions: Behavioral: Quality Training
- Goal Training Group (Active Comparator)
  Interventions: Behavioral: Goal Training

INTERVENTIONS:
Behavioral: Quality Training — Participants will engage in piano playing tasks using their affected hand and fingers. The training focuses on specific aspects of finger movement, and participants will receive feedback related to their playing. They will wear a wrist brace for support, and their hand and arm positions will be monitored to ensure proper technique.
  Arms: Quality Training Group
Behavioral: Goal Training — Participants will engage in piano playing tasks using their affected hand and fingers. The training emphasizes learning to play and producing music. Feedback will be provided on various aspects of performance such as speed and accuracy, but specific details about finger movement or technique will not be given. The use of a wrist brace and monitoring of hand and arm positions will be consistent with standard practice.
  Arms: Goal Training Group

SUMMARY:
The goal of this clinical trial is to compare two rehabilitation methods to improve finger movements in people who have had a stroke. The main question it aims to answer is which of these two training methods leads to the most improvement:

1. Teaching people to reach their movement goals using any strategies they like.
2. Teaching people to improve their movement technique and avoid compensatory strategies.

There is no one-size-fits-all approach. The second goal is to find out who might benefit more from each method. Some people with stroke may rely on compensatory strategies due to severe impairment, while others with milder strokes might benefit more from techniques that enhance movement quality.

The third goal is to take pictures of the brain to see how it changes with each method. This will help researchers understand how the brain adapts after a stroke and could lead to treatments that target the brain directly.

Participants will:

1. Visit the lab for clinical and research assessments on weeks 1, 4, 5, and 15.
2. Complete 10 days of piano training.
3. Undergo magnetic resonance imaging (MRI) scans twice, once in week 1 and once in week 4.

DETAILED DESCRIPTION:
Forty participants with sub-acute (6 months - 2 years) stroke will be recruited in this multi-site trial taking place in Toronto and Montreal. Participants will need to be able to perform active finger movements. Each site will recruit and randomize participants into one of two training groups. Training will consist of:

1. One group will focus on improving the quality of their movements while playing music on a digital piano.
2. The other group will focus on achieving their movement goals while playing playing music on a digital piano.

Participation in this study will involve 14 visits, each taking place on a separate day.

Piano training consists of 20 hours total, spread over 2 hours per day for 5 days across 2 weeks. Each participant will receive one-on-one and/or group instruction from a Music Therapist with expertise in Neurologic Music Therapy and piano instruction. Exercises will include pressing single keys and multiple keys with different fingers, holding down certain keys while pressing others, and playing melodies and chords with all five fingers, involving various coordination patterns, rhythms, and speeds.

Assessments will be conducted at four timepoints: Baseline, Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months). Participants will undergo validated clinical assessments to evaluate their ability to move and feel their arm, hand, and fingers, as well as for assessor to understand how the stroke has affected them overall. Some of these tests are routinely used by physical therapists and other rehabilitation professionals who work with people living with stroke. For other types of tests, sensors will be placed on their arm, hand, and fingers. These sensors do not emit anything; they will simply record their movements.

Kinetic and kinematic measures will assess finger forces, grip strength, and pinch strength. Magnetic resonance imaging (MRI) scans at Baseline and Post-training-1 will be taken to quantify structure and function of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosis of first time unilateral ischemic or hemorrhagic
* Stroke occurrence: > 6 months and < 2 years
* Able to perform active finger movements (Chedoke-McMaster (CM) Impairment Inventory of the Hand, Stage ≥ 3)

Exclusion Criteria:

* History of developmental, neurological, or major psychiatric disorders
* Cognitive deficits (< 23/30 Montreal Cognitive Assessment)
* Apraxia (<2SD mean Waterloo Apraxia test)
* Neglect (> 40/100, Sunnybrook Neglect Assessment Procedure)
* Cerebellar stroke
* Musculoskeletal injury affecting motor performance
* Inability to sit in a chair and perform exercises for sustained periods
* Contraindications to MRI

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Finger Individuation: Force | Pre-training (baseline), Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months)
  The Finger Individuation - Force is a measure of how well a finger is able to exert force without the other fingers exerting force. This measure has been used to study finger movements in healthy individuals, pianists, and stroke survivors. This task will use a custom device to measure finger movements in all digits of both hands. The forearm will be placed on a table with the wrist in a neutral position and secured to prevent other movements. The device will support the palm and measure the force each finger produces using sensors under each fingertip. The investigators will determine participants' maximum finger force. Then, participants will practice producing forces at 20%, 40%, 60%, and 80% of this maximum for each finger while keeping the others still. They will see a visual target for the required force and get feedback on their performance.
Finger Individuation: Joint Angular Excursion | Pre-training (baseline), Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months).
  The Finger Individuation - Joint Angular Excursion is a measure of how well a finger is able to bend or straighten while the other fingers remain stationary. The angle being measured in this task is the degree of flexion and extension at the finger joints. Specifically, it tracks the movement at the metacarpophalangeal (MCP) joint (i.e., the joint where the finger meets the hand), and proximal interphalangeal (PIP) joint (i.e., joint between the first and second finger bones). Infrared markers will be placed on the metacarpal MCP and PIP joints to track finger movement using two 3-camera Optotrak Certus motion capture systems.

SECONDARY OUTCOMES:
Fugl Meyer Upper Limb assessment (FM-UL) | Pre-training (baseline), Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months).
  The FM-UL assessment assesses the sensorimotor impairment in individuals who have had stroke. It assesses movements, coordination, and reflexes.
Action Research Arm Test (ARAT) | Pre-training (baseline), Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months).
  The ARAT is a 19-item assessment designed to evaluate upper extremity motor activity. It measures how well individuals can perform specific arm and hand tasks, focusing on four main areas: grasp, grip, pinch, and gross movement.
Nine-Hole Peg Test (9-HPT) | Pre-training (baseline), Post-training-1 (day 3), Post-training-2 (day 7), and Follow-up (3 months).
  The 9-HPT is a standardized, quantitative assessment designed to evaluate finger dexterity. In this test, participants are required to pick up pegs from a container one at a time and place them into holes on a pegboard as quickly as possible.
MRI: Neural activation and connectivity in ipsilesional and contralesional motor cortex | Baseline and Post-training-1 (day 3)
  The investigators will examine how various areas of the brain function and interact, with a focus on the regions that control movement. They will specifically assess both the injured side of the brain (ipsilesional) and the uninjured side (contralesional) to observe how each responds during tasks.
MRI: White matter integrity in corticospinal, reticulospinal and rubrospinal tracts | Baseline and Post-training-1 (day 3)
  The investigators will evaluate the condition of specific brain pathways involved in transmitting signals to participants' muscles, including the corticospinal, reticulospinal, and rubrospinal tracts.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce L Chen, PhD, Principal Investigator — University of Toronto: Faculty of Kinesiology & Physical Education
Locations (5):
- Canada (5):
  - University of Toronto, Toronto, Ontario
  - Jewish Rehabilitation Hospital, Laval, Quebec
  - University Institute for Physical Impairment Rehabilitation of Montreal (IURDPM), Montreal, Quebec
  - Lethbridge-Layton-Mackay Rehabilitation Center, Montreal, Quebec
  - Jewish General Hopsital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposals should be directed to JOYCELYNN.CHEN@UTORONTO.CA. To gain access, data requestors will need to sign a data transfer agreement.